CLINICAL TRIAL: NCT05081882
Title: Reducing Tobacco-associated Lung Cancer Risk: A Randomized Clinical Trial of AB-free Kava
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kava; OCR40933 (Other: University of Florida); IRB202101885 (Other: University of Florida IRB-01)
Record Dates: First submitted 2021-09-21; First posted 2021-10-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Smoking
Keywords: tobacco dependence; smoking cessation; kava
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Kava Intervention (Experimental)
  Interventions: Drug: Kava
- Placebo Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kava — Participants on this arm will take one kava capsule (each capsule contains 75 mg of kavalactones) orally three times daily for 28 days.
  Arms: Kava Intervention
Drug: Placebo — Participants on this arm will take one placebo capsule orally three times daily for 28 days.
  Arms: Placebo Control

SUMMARY:
Tobacco use is the leading cause of many preventable diseases, particularly lung cancer. Based on the national cancer data in 2020, Florida has the highest lung cancer incidence (18,150 cases) with the most deaths (10,580 deaths) among all the states in the United States. Unfortunately, around 16% of adults in Florida continue to smoke cigarettes due to its addictive nature and the limited success of current cessation strategies. Therefore, there is an unmet and urgent need for novel interventions to improve the success of tobacco cessation. If such an intervention can reduce tobacco-associated lung carcinogenesis, that will be more desirable. The ultimate goal of this study is to develop a safe and effective kava-based intervention to enable tobacco cessation and reduce lung cancer risk, which will improve the health of Floridians.

This study will evaluate the compliance with a daily kava regimen among active smokers who have no intention to quit smoking. This study will also investigate whether kava use can reduce tobacco use and dependence, as well as tobacco-associated lung carcinogenesis.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 21 years or above
* self-reported smoking at least 5 cigarettes/day for the past year with no intention to quit at time of screening visit
* expired carbon monoxide level of more than 8 ppm at recruitment
* willingness to participate in the proposed study, as indicated by signed informed consent
* access to a functional telephone
* expected presence in the study's geographical area for the next 4 months
* not currently enrolled in any smoking cessation programs per self-report
* female subjects of childbearing potential will be required to practice acceptable methods of birth control (the acceptable methods of birth control include birth control pills, Birth Control Shot, Birth Control Implant, Intrauterine Device [IUD], Diaphragm, and cervical cap)

Exclusion Criteria:

* history of active cancer (other than non-melanoma skin cancer) within the past 2 years
* diagnosed with liver dysfunction or with previous liver diseases
* levels of alanine transaminase, aspartate transaminase, alkaline phosphatase, or total bilirubin over limit of normal range at prescreen
* inability to refrain from acetaminophen, alcohol (no more than one drink daily via self-report)
* are pregnant or nursing (lactating) or of childbearing age planning to become pregnant or unwilling to use adequate contraception during the study
* participant answered "Yes" to any of the ASQ questions 1 through 3, or refuses to answer all of the questions. If subject answers 'Yes' to question 4 but the most recent suicide attempt took place more than12 months from screening visit then subject is still eligible.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Subject Compliance with Intervention | 4 weeks
  Evaluate subject compliance with the kava intervention, as measured by participant reported number of missed doses
Subject Compliance with Intervention | 4 weeks
  Evaluate subject compliance with the kava intervention, as measured by detection of dihydromethysticin in participant urine

SECONDARY OUTCOMES:
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by participant reported number of cigarettes smoked
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Fagerström Test for Nicotine Dependence (FTND)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Modified Cigarette Evaluation Questionnaire (mCEQ)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by the Brief Questionnaire on Smoking Urges (QSU-Brief)
Tobacco cessation | 12 weeks
  Examine whether kava has the potential to help facilitate tobacco cessation, as measured by urinary total nicotine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Xing C, Malaty J, Malham MB, Nehme AMA, Freeman B, Huo Z, Firpi-Morrel R, Salloum RG. Reducing tobacco-associated lung cancer risk: a study protocol for a randomized clinical trial of AB-free kava. Trials. 2023 Jan 18;24(1):36. doi: 10.1186/s13063-023-07081-x. PMID 36653872